CLINICAL TRIAL: NCT05803941
Title: A Phase IV, Post-Authorization Safety Study to Investigate the Long-Term Safety of Lutetium (177Lu) Vipivotide Tetraxetan in Adult Participants With Prostate Cancer
Brief Title: Long-Term Safety of Lutetium (177Lu) Vipivotide Tetraxetan in Participants With Prostate Cancer
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CAAA617A12402; 2023-503208-94-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2023-03-27; First posted 2023-04-07 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Long-Term Safety Follow-Up; 177Lu-PSMA-617; [177Lu]Lu-PSMA-617; lutetium (177Lu) vipivotide tetraxetan; AAA617; parent treatment study
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Lutetium; Lutetium-177; Pluvicto

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single arm (Other): Participants will be followed until death, lost to follow-up, or up to 10 years from first dose of AAA617, whichever occurs first.
  There will be no study treatment administered to participants while participating in this study.
  Interventions: Drug: AAA617

INTERVENTIONS:
Drug: AAA617 — Long-term follow-up (LTFU) safety study of adult participants with prostate cancer that have received at least one dose of AAA617 from parent interventional Novartis sponsored clinical trials.
  Other Names: lutetium (177Lu) vipivotide tetraxetan; [177Lu]Lu-PSMA-617; 177Lu-PSMA-617

SUMMARY:
The purpose of this post-marketing study is to further characterize the long-term outcome of known or potential risks of lutetium (177Lu) vipivotide tetraxetan also known as [177Lu]Lu-PSMA-617 or 177Lu-PSMA-617 and hereinafter referred to as AAA617. The study also seeks to further characterize (as possible) any other AAA617 causally related serious adverse event(s) in the long-term in adults with prostate cancer who received at least one dose of AAA617 from interventional, Phase I-IV Novartis sponsored clinical trials.

DETAILED DESCRIPTION:
This is a global, prospective, multi-center, long-term follow-up (LTFU) safety study of adult participants with prostate cancer that have received at least one dose of AAA617 from interventional, Phase I-IV Novartis sponsored clinical trials.

There will be no study treatment administered to participants in this study. Participants will have visits every 6-8 months for monitoring of selected AEs and laboratory parameters. The study periods include a Baseline and Follow-up Period (up to 10 years after first dose of AAA617 in parent treatment study).

Participants should enroll into the LTFU study after parent treatment study requirements are fulfilled (refer to the parent treatment study protocol for requirements, including any additional requirements after participant enters this LTFU safety study).

The schedule of activities for this LTFU study is designed to start from date of informed consent for this LTFU study. Participants should be followed every 6 to 8 months for up to a total of 10 years starting from first dose of AAA617 in the parent treatment study. Participants entering the LTFU study will have already completed a variable portion of the required 10-year follow-up within the parent treatment study. The specific number of visits required in this LTFU study will depend upon the time of enrollment into this LTFU study following the first dose of AAA617 in the parent treatment study.

The total number of participants to be enrolled and the duration of this LTFU study will depend upon the total number treated in the parent treatment studies and their duration.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent must be obtained prior to participation in the study
* Must have received at least one dose of AAA617 within an interventional, Phase I-IV Novartis sponsored clinical trial in prostate cancer and have fulfilled the trial's requirements that allows them to participate in this study.

Exclusion Criteria:

- Inability to complete the needed investigational examinations due to any reason.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer
Enrollment: 700 (Estimated)
Dates: Start 2023-08-14 (Actual); Primary Completion 2033-07-20 (Estimated); Study Completion 2033-07-21 (Estimated)

PRIMARY OUTCOMES:
Number and percentage of participants with selected Adverse Events (AEs) and Serious Adverse Events (SAEs) | every visit up to 10 years after 1st dose of AAA617 received in parent treatment study
  Selected adverse events (AEs) include xerostomia, xerophtalmia, myelosupression, renal toxicity and second primary malignancy and their complication. Only SAEs considered causally related to previous treatment with AAA617 will be considered.

SECONDARY OUTCOMES:
Number and percentage of participants who have died | every visit up to 10 years after 1st dose of AAA617 received in parent treatment study
  The number and percentage of participants who die during the long-term follow-up will be summarized.
Absorbed radiation dose in kidney or other selected organs and number of AEs | every visit up to 10 years after 1st dose of AAA617 received in parent treatment study
  Correlation between absorbed radiation dose in kidney or selected organs and safety of AAA617 for participants with dosimetry estimates collected in the parent treatment study.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (49):
- United States (24):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - St. Joseph Hospital, Orange, California
  - Providence Saint Johns Health Ctr, Santa Monica, California
  - University of Colorado, Aurora, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - VA Medical Center, Washington D.C., District of Columbia
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - University Cancer and Blood Center LLC, Athens, Georgia
  - Parkview Research Center, Fort Wayne, Indiana
  - Tulane Cancer Center, New Orleans, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Corewell Health William Beaum Hosp, Royal Oak, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - University of Mississippi Med Ctr, Jackson, Mississippi
  - Wash U School of Medicine, St Louis, Missouri
  - Urology Cancer Center PC, Omaha, Nebraska
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Univ of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Univ of Texas Southwest Med Center, Dallas, Texas
  - UT Health Science Center, Houston, Texas
  - Onco Hemato Asso of SE Virginia, Roanoke, Virginia
- Austria (2):
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Vienna
- Novartis Investigative Site, Ghent, Belgium
- Novartis Investigative Site, Montreal, Quebec, Canada
- Czechia (2):
  - Novartis Investigative Site, Olomouc
  - Novartis Investigative Site, Prague
- Novartis Investigative Site, Lyon, France
- Germany (3):
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Rostock
- Netherlands (3):
  - Novartis Investigative Site, Delft
  - Novartis Investigative Site, Maastricht
  - Novartis Investigative Site, Nijmegen
- Spain (5):
  - Novartis Investigative Site, Sabadell, Barcelona
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Valencia
- Sweden (2):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Stockholm
- United Kingdom (5):
  - Novartis Investigative Site, Sutton, Surrey
  - Novartis Investigative Site, Barnet
  - Novartis Investigative Site, Cambridge
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, Middlesbrough

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.